CLINICAL TRIAL: NCT00825929
Title: Study on Pharmacokinetics of Newly Developed ANtiretroviral Agents in HIV-infected pregNAnt Women (PANNA)
Brief Title: Pharmacokinetics of Antiretroviral Agents in HIV-infected Pregnant Women.
Acronym: PANNA
Status: Recruiting | Type: Observational
Sponsor: Radboud University Medical Center (Other)
Collaborators: PENTA Foundation (Network); Merck Sharp & Dohme LLC (Industry); Bristol-Myers Squibb (Industry); Janssen Pharmaceutica (Industry); ViiV Healthcare (Industry); Gilead Sciences (Industry)
Responsible Party: Sponsor
Other Study IDs: UMCN-AKF 08.02
Record Dates: First submitted 2009-01-19; First posted 2009-01-21 (Estimated); Last update posted 2025-01-13 (Actual); Status verified 2025-01

CONDITIONS: HIV Infections
Keywords: pharmacokinetics; pregnancy; antiretrovirals; neonates; HIV; treatment experienced
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma samples will be collected in Week 33 of the pregnancy and at 4-6 weeks after delivery. At the following time points T=0 (prior to dosing), and T=1, 2, 3, 4, 6, 8, 12 and 24h (24h sample only in case of QD regimen) post-dosing (8 or 9 samples).
  In case the infant needs post-exposure prophylaxis with at least one of the agents sparse PK sampling is optional.
  If the mother decides to breastfeed, also breast milk samples at 2, 4, 6, 12 and 24 hours after dosing will be collected on the postpartum PK day.
  For CAB/RPV:
  Maternal PK curve after the injection from 24 weeks gestational age and after first or second injection postpartum: one sample prior to injection, and at day 3, 7, 28 and 56 (in case of 2 monthly injections).
  If the mother decides to breastfeed, also breast milk samples at the same postpartum timepoints and one infant blood sample (extra consent) will be collected.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Treated with one of the antiretroviral agents under study, PK parameters during pregnancy will be compared with PK parameters after pregnancy (within the same woman)

SUMMARY:
Due to the potential for pregnancy-induced changes in the pharmacokinetics of medication, one cannot assume that the currently licensed doses of the medication to be tested under this protocol lead to adequate exposure in an HIV-infected pregnant woman. For the agents under study no or limited pharmacokinetic data during pregnancy are available. As the changes in pharmacokinetics during pregnancy are most prominent in the third trimester a pharmacokinetic curve will be recorded in the third trimester after attaining steady state.

DETAILED DESCRIPTION:
The following agents will be studied:

Etravirine, Intelence, TMC125; Emtricitabine, Emtriva or FTC; Tenofovir, Viread, TDF; Atazanavir, Reyataz; Fosamprenavir, Telzir, FPV; Darunavir, Prezista, TMC114; Tipranavir, Aptivus, TPV; Indinavir, Crixivan; abacavir; raltegravir, Isentress; Enfuvirtide, Fuzeon; Maraviroc, Celsentri; dolutegravir; elvitegravir/cobicistat; rilpivirine, TAF, darunavir/cobicistat; doravirine; bictegravir; cabotegravir/rilpivirine long acting injectables

ELIGIBILITY:
Inclusion Criteria:

1. HIV-infected as documented by positive HIV antibody test and confirmed by an antigen test.
2. Subject is at least 18 years of age at screening.
3. Subject is able and willing to sign the Informed Consent Form prior to screening evaluations.
4. Treated with a cART regimen containing at least one agent which is mentioned in Appendix 1; this agent has been taken for at least 2 weeks before the day of first PK curve evaluation.
5. Subject is pregnant
6. Subject is able to adhere to food intake recommendations, if applicable.

Exclusion Criteria:

1. Relevant history or current condition that might interfere with drug absorption, distribution, metabolism or excretion.
2. Inability to understand the nature and extent of the study and the procedures required.
3. Presence of grade III/IV anemia (i.e. Hb <4.6 mmol/L or <7.4 g/dL).
4. Using oral cabotegravir/rilpivirine.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HIV-infected pregnant women using at least one of the following antiretroverial agents: Etravirine, Intelence, TMC125; Emtricitabine, Emtriva or FTC; Tenofovir, Viread, TDF; Atazanavir, Reyataz; Fosamprenavir, Telzir, FPV; Darunavir, Prezista, TMC114; Tipranavir, Aptivus, TPV; Indinavir, Crixivan; abacavir; raltegravir, Isentress; Enfuvirtide, Fuzeon; Maraviroc, Celsentri; dolutegravir; elvitegravir/cobicistat; rilpivirine, TAF, darunavir/cobicistat; doravirine; bictegravir; cabotegravir/rilpivirine LA
Sampling Method: Non-Probability Sample
Enrollment: 176 (Estimated)
Dates: Start 2009-02; Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Plasma concentrations of the compounds during pregnancy compared to the concentrations after delivery | PK curve in Week 33 of pregnancy and 4-6 weeks after delivery

SECONDARY OUTCOMES:
Pharmacokinetics in the neonate, in case of post-exposure prophylaxis with one of the agents under study. | Week 1, 3 and between 4 and 6
Safety of antiretrovirals during pregnancy | GA Week 33 until end of trial
viral load response and prevention of mother to child transmission of the virus | GA Week 3 and at delivery

CONTACTS AND LOCATIONS:
Overall Officials: David M Burger, PharmD PhD, Principal Investigator — Radboud University Medical Centre Nijmegen
Locations (21):
- Saint-Pierre University Hospital; Department of Infectious Diseases, Brussels, Belgium
- Germany (5):
  - CHARITÉ Berlin, Berlin
  - University of Bonn, Bonn
  - University of Cologne, Cologne
  - Johann Wolfgang Goethe-Universität, Frankfurt am Main
  - University München, München
- Ireland (2):
  - Mater Hospital and UCD, Dublin
  - St James's Hospital Dublin, Dublin
- IRCSS, Rome, Italy
- Netherlands (4):
  - AMC, Amsterdam
  - Radboud University Nijmegen Medical Centre, Nijmegen
  - Erasmus Medical Center Rotterdam, Rotterdam
  - St Elisabeth hospital, Tilburg
- Spain (2):
  - Hospital Universitari Germans Trias i Pujol, Badalona, Badalona
  - Hospital Universitario Virgen de las Nieves Granada; Médico Adjunto del Servicio de Medicina Interna, Granada
- United Kingdom (6):
  - Brighton and Sussex University Hospitals NHS Trust, Brighton
  - C&W Hospital, London, London
  - North Middlesex Hospital, London
  - St Mary's Hospital, London, London
  - St Thomas Hospital, London
  - St. George's Hospital, London, London

REFERENCES:
- [Result] Colbers AP, Hawkins DA, Gingelmaier A, Kabeya K, Rockstroh JK, Wyen C, Weizsacker K, Sadiq ST, Ivanovic J, Giaquinto C, Taylor GP, Molto J, Burger DM; PANNA network. The pharmacokinetics, safety and efficacy of tenofovir and emtricitabine in HIV-1-infected pregnant women. AIDS. 2013 Mar 13;27(5):739-48. doi: 10.1097/QAD.0b013e32835c208b. PMID 23169329
- [Result] Colbers A, Gingelmaier A, van der Ende M, Rijnders B, Burger D. Pharmacokinetics, safety and transplacental passage of rilpivirine in pregnancy: two cases. AIDS. 2014 Jan 14;28(2):288-90. doi: 10.1097/QAD.0000000000000100. No abstract available. PMID 24413315
- [Result] Bollen P, Freriksen J, Konopnicki D, Weizsacker K, Hidalgo Tenorio C, Molto J, Taylor G, Alba-Alejandre I, van Crevel R, Colbers A, Burger D; Pharmacokinetics of ANtiretroviral agents in HIV-infected pregNAnt women Network. The Effect of Pregnancy on the Pharmacokinetics of Total and Unbound Dolutegravir and Its Main Metabolite in Women Living With Human Immunodeficiency Virus. Clin Infect Dis. 2021 Jan 23;72(1):121-127. doi: 10.1093/cid/ciaa006. PMID 32103260
- [Derived] Overbeek JK, van Erp NP, Burger DM, den Broeder AA, Koolen SLW, Huitema ADR, Ter Heine R. Population Pharmacokinetics of Cobicistat and its Effect on the Pharmacokinetics of the Anticancer Drug Olaparib. Clin Pharmacokinet. 2025 Mar;64(3):425-435. doi: 10.1007/s40262-025-01480-w. Epub 2025 Feb 5. PMID 39909979
- [Derived] Bukkems V, Necsoi C, Tenorio CH, Garcia C, Rockstroh J, Schwarze-Zander C, Lambert JS, Burger D, Konopnicki D, Colbers A. Clinically Significant Lower Elvitegravir Exposure During the Third Trimester of Pregnant Patients Living With Human Immunodeficiency Virus: Data From the Pharmacokinetics of ANtiretroviral agents in HIV-infected pregNAnt women (PANNA) Network. Clin Infect Dis. 2020 Dec 17;71(10):e714-e717. doi: 10.1093/cid/ciaa488. PMID 32330231
- [Derived] Kreitchmann R, Schalkwijk S, Best B, Wang J, Colbers A, Stek A, Shapiro D, Cressey T, Mirochnick M, Burger D. Efavirenz pharmacokinetics during pregnancy and infant washout. Antivir Ther. 2019;24(2):95-103. doi: 10.3851/IMP3283. PMID 30530925
- [Derived] Schalkwijk S, Colbers A, Konopnicki D, Gingelmaier A, Lambert J, van der Ende M, Molto J, Burger D; Pharmacokinetics of newly developed antiretroviral agents in HIV-infected pregnant women (PANNA) Network. Lowered Rilpivirine Exposure During the Third Trimester of Pregnancy in Human Immunodeficiency Virus Type 1-Infected Women. Clin Infect Dis. 2017 Oct 15;65(8):1335-1341. doi: 10.1093/cid/cix534. PMID 28595298
- [Derived] Mulligan N, Schalkwijk S, Best BM, Colbers A, Wang J, Capparelli EV, Molto J, Stek AM, Taylor G, Smith E, Hidalgo Tenorio C, Chakhtoura N, van Kasteren M, Fletcher CV, Mirochnick M, Burger D. Etravirine Pharmacokinetics in HIV-Infected Pregnant Women. Front Pharmacol. 2016 Aug 4;7:239. doi: 10.3389/fphar.2016.00239. eCollection 2016. PMID 27540363
- [Derived] Colbers A, Best B, Schalkwijk S, Wang J, Stek A, Hidalgo Tenorio C, Hawkins D, Taylor G, Kreitchmann R, Burchett S, Haberl A, Kabeya K, van Kasteren M, Smith E, Capparelli E, Burger D, Mirochnick M; PANNA Network and the IMPAACT 1026 Study Team. Maraviroc Pharmacokinetics in HIV-1-Infected Pregnant Women. Clin Infect Dis. 2015 Nov 15;61(10):1582-9. doi: 10.1093/cid/civ587. Epub 2015 Jul 22. PMID 26202768
- [Derived] Blonk MI, Colbers AP, Hidalgo-Tenorio C, Kabeya K, Weizsacker K, Haberl AE, Molto J, Hawkins DA, van der Ende ME, Gingelmaier A, Taylor GP, Ivanovic J, Giaquinto C, Burger DM; Pharmacokinetics of Newly Developed Antiretroviral Agents in HIV-Infected Pregnant Women PANNA Network; PANNA Network. Raltegravir in HIV-1-Infected Pregnant Women: Pharmacokinetics, Safety, and Efficacy. Clin Infect Dis. 2015 Sep 1;61(5):809-16. doi: 10.1093/cid/civ366. Epub 2015 May 5. PMID 25944344
- [Derived] Colbers A, Molto J, Ivanovic J, Kabeya K, Hawkins D, Gingelmaier A, Taylor G, Weizsacker K, Sadiq ST, Van der Ende M, Giaquinto C, Burger D; PANNA Network. Pharmacokinetics of total and unbound darunavir in HIV-1-infected pregnant women. J Antimicrob Chemother. 2015 Feb;70(2):534-42. doi: 10.1093/jac/dku400. Epub 2014 Oct 17. PMID 25326090
- [Derived] Colbers A, Hawkins D, Hidalgo-Tenorio C, van der Ende M, Gingelmaier A, Weizsacker K, Kabeya K, Taylor G, Rockstroh J, Lambert J, Molto J, Wyen C, Sadiq ST, Ivanovic J, Giaquinto C, Burger D; PANNA network. Atazanavir exposure is effective during pregnancy regardless of tenofovir use. Antivir Ther. 2015;20(1):57-64. doi: 10.3851/IMP2820. Epub 2014 Jul 3. PMID 24992294
- See also: PANNA study website — http://www.pannastudy.com